CLINICAL TRIAL: NCT01660984
Title: Longitudinal Assessment and Natural History Study of Children and Adults With MEN2A or MEN2B With or Without Medullary Thyroid Carcinoma
Brief Title: Natural History Study of Children and Adults With Medullary Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120178; 12-C-0178
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-10-16

CONDITIONS: Medullary Thyroid Cancer
Keywords: Thyroid Tumor; Multiple Endocrine Neoplasia 2; Pheochromocytoma; RET Mutations; Natural History
MeSH Terms: conditions — Carcinoma, Medullary; Thyroid Neoplasms; Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents/caregivers: Parents or caregivers of study patients to assess their psychosocial experiences and needs.
- Patients: Children and adults with MTC and MEN2B, other non-tumor manifestations of MEN2, and patients with MEN2 who do not demonstrate MTC. Characterize the biology and manifestations of their disease.

SUMMARY:
Background:

- Medullary thyroid cancer (MTC) is a rare cancer of the thyroid gland. In children and adults, it is often part of a condition called Multiple Endocrine Neoplasia 2 (MEN2). MEN2 is usually caused by a genetic mutation, and it can cause a number of problems in addition to MTC. These problems include adrenal gland tumors, hormone changes, and problems with the bones and other organs. Not much is known about how MTC develops over time, especially in people with MEN2. Researchers want to study MTC in children and adults and see how it affects their growth and development.

Objectives:

- To study how medullary thyroid cancer affects children and adults over time.

Eligibility:

- Children and adults who have medullary thyroid cancer.

Design:

* Participants will be screened with a brief physical exam and medical history. Blood and tissue samples will be collected to see whether participants have the MEN2 genetic mutation.
* Treatment will not be provided as part of this study. However, participants will be receiving standard care for MTC. They may be eligible for other clinical trials at the National Institutes of Health.
* Participants will have regular study visits every 6 to 12 months to evaluate their MTC and any treatment. Blood tests, imaging studies, and other tests may be performed as needed to monitor the disease.
* Participants and their parents/guardians will also complete questionnaires about their health and emotions during the study.

DETAILED DESCRIPTION:
Background:

* Medullary Thyroid Carcinoma (MTC) is a calcitonin producing tumor arising from the parafollicular C cells of thyroid. In children and adults, MTC is usually seen in association with Multiple Endocrine Neoplasia (MEN) 2A and 2B, which are rare cancer syndromes resulting from germline mutations of Rearranged during Transfection (RET) proto-oncogene. MTC develops in virtually all patients with MEN 2, and is the leading cause of death in these patients. Patients with MEN 2 may have other characteristic manifestations such as pheochromocytoma and hyperparathyroidism in MEN 2A and pheochromocytoma, ganglioneuromatosis, and skeletal deformities in MEN 2B.
* Complete surgical resection is the only current curative treatment for MTC, and the tumor is unresponsive to standard chemotherapy and conventional doses of radiation therapy. However, more than half the patients present with advanced or metastatic disease and cannot be cured surgically. Novel agents are currently under investigation for treatment of MTC, and vandetanib, an oral RET and receptor tyrosine kinase (RTK) inhibitor was recently approved by the FDA for adults with advanced or metastatic MTC. Vandetanib also has activity in children with hereditary MTC.
* However, complete responses to RTKs have not been observed, and some patients develop resistance to the treatment with RET and RTK inhibitors or have primary refractory disease. The natural history of MTC, particularly in patients with MEN 2, the molecular pathways involved in tumorigenesis, and the development of resistance to targeted therapies are not well understood.

Objectives:

-The overall objective of this longitudinal study is to develop a better understanding of the biology and natural history of MEN2 with or without MTC, particularly in children and adults with MEN 2A and 2B, as well as study non-tumor manifestations of MEN 2. This will hopefully allow for developing more effective treatment interventions for tumor and non-tumor related manifestations, and more sensitive endpoints in clinical trials.

Eligibility:

* Patients, must have histologically or cytologically confirmed MTC, confirmed by the Laboratory of Pathology, NCI or who have MEN2 (regardless of MTC status).
* Parent or primary caregiver of patient participant (<= 21)
* Participants may be undergoing standard care or receiving treatment on a clinical trial while participating in this study.

Design:

This study will allow for longitudinal evaluations of MTC and MEN2 and non-tumor related manifestations of MEN 2A and 2B in children and adults. Evaluations will consist of the following (summarized):

1. Clinical and radiological evaluations
2. Detailed pathologic and molecular analysis of tumor specimens will be performed, including immunohistochemistry (IHC), comparative genomic hybridization (CGH), and genome sequencing. CGH and genome sequencing will be performd with co-enrollment on protocol 10-C-0086 Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENTS:
* Patients must have histologically or cytologically confirmed MTC, confirmed by the Laboratory of Pathology, NCI OR Confirmation of MEN2A or MEN2B diagnosis, regardless of presence of MTC.
* Performance Status: Ability to travel to the NIH and to undergo evaluations to be performed on this protocol.
* Informed Consent: Ability of patient or their legal guardian (if the patient is <18 years old) to understand and willing to sign a written informed consent document.
* Prior and current therapy: For the purpose of this study subjects who have not previously received medical or surgical treatment, patients, who have previously received medical or surgical treatment, and subjects who are currently receiving medical treatment and/or radiation for MEN 2 related manifestation(s) will be eligible. Prior and current treatment for MEN 2 related manifestations will be recorded at trial entry and throughout the study.
* Patients must have a primary care provider (for example a primary oncologist or endocrinologist) who can provide and coordinate the medical care for the patient.

EXCLUSION CRITERIA FOR PATIENTS:

-In the opinion of the investigator the patient is not able to return for follow-up visits or obtain required follow-up studies.

Inclusion Criteria for Parents or Primary Caregivers

* Must be a parent or primary caregiver of a patient (< 21) who has a histologically or cytologically confirmed MTC or who have MEN2 (regardless of MTC status).
* Ability to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA FOR PARENTS OR PRIMARY CAREGIVERS: None

Min Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed MTC, confirmed by the Laboratory of Pathology, NCI, or confirmed MEN2A or MEN2B diagnosis, regardless of presence of MTC. Parents or caregivers of the enrolled patients will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Estimated)
Dates: Start 2012-07-30 (Actual)

PRIMARY OUTCOMES:
Study growth rate of primary and metastatic tumor lesions | 5 years
  Characterized features will be described and presented.
Study molecular pathways altered in MTC | 5 years
  Characterized features will be described and presented.

SECONDARY OUTCOMES:
Describe the non-tumor related manifestations of MEN 2 | 5 years
  Describe the non-tumor related manifestations of MEN 2
Investigate the psychosocial experiences | 5 years
  Investigate the psychosocial experiences

CONTACTS AND LOCATIONS:
Overall Officials: John W Glod, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Li I, Hartley IR, Klubo-Gwiedzdzinska J, Reynolds JC, Thomas BJ, Hogan J, Enyew MM, Dombi E, Ling A, Akshintala S, Venzon DJ, Del Rivero J, Collins M, Glod JW. Fracture Risk in Pediatric Patients With MEN2B. J Clin Endocrinol Metab. 2022 Nov 25;107(12):e4371-e4378. doi: 10.1210/clinem/dgac500. PMID 36056624
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-C-0178.html